CLINICAL TRIAL: NCT06096987
Title: Examining the Effects of MyChart Peer Education on Adolescent Health Literacy and Engagement With Personal Health Information
Brief Title: Teen-to-Teen Videos to Improve Electronic Medical Record Portal Knowledge and Personal Health Information Engagement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huang, Jeannie, M.D. (Individual)
Collaborators: North American Society for Pediatric Gastroenterology Hepatology and Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 804613
Record Dates: First submitted 2023-09-21; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic medical record portal video group (Experimental): Assigned to receive videos regarding electronic medical record portals and information shared in electronic medical record portals
  Interventions: Other: Electronic medical record portal videos
- General adolescent health video group (Active Comparator): Assigned to receive videos regarding general adolescent health issues
  Interventions: Other: General adolescent health videos

INTERVENTIONS:
Other: Electronic medical record portal videos — Teen to teen videos reviewing information about electronic medical record portals and information shared in electronic medical record portals.
  Arms: Electronic medical record portal video group
Other: General adolescent health videos — Teen to teen videos reviewing information about general adolescent health issues.
  Arms: General adolescent health video group

SUMMARY:
The goal of this clinical trial is to compare whether videos help teens better understand medical topics. The main questions answered in this trial are:

1. whether videos can improve teen knowledge about electronic medical record portals
2. whether videos can improve teen knowledge about general health issues

Participants will answer surveys and watch videos as part of this study.

DETAILED DESCRIPTION:
Investigators performed a randomized controlled trial of education videos addressing one of two topics: A) electronic medical record portals and information shared therein and B) general adolescent health issues among adolescents and young adults with inflammatory bowel diseases. Investigators evaluated the efficacy of each in increasing participant knowledge in that arena.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Inflammatory Bowel Disease
* English proficient

Exclusion Criteria:

- Unable to give consent

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Electronic medical record (EMR) portal knowledge assessment | Baseline and Immediately after video watching (all done SAME DAY - 1 day)
  12 questions about EMR portals and information shared via EMR portals to measure participants' knowledge about EMR portals. Measured as percent correct out of 100% with higher correct indication greater knowledge.
General adolescent health knowledge assessment | Baseline and Immediately after video watching (all done SAME DAY - 1 day)
  12 Questions about general adolescent health issues to measure participants' knowledge in these areas. Measured as percent correct out of 100% with higher correct indication greater knowledge.

SECONDARY OUTCOMES:
Short Test of Functional Health Literacy in Adults | At baseline
  An adult health literacy measure consisting of 36 comprehension questions and 4 numeric calculations scored on a scale of 0-36 with a score of 23 set as the threshold for adequate health literacy

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Huang, MD, MPH, Principal Investigator — University of California San Diego/Rady Children's Hospital
Locations (1):
- Rady Children's Hospital, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No